CLINICAL TRIAL: NCT01523795
Title: PRESENCE 2: Predicting Sedentary Entertainment Choices and Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10-1415
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Obesity; Physical Activity
Keywords: Energy intake; Video games; Television; Physical activity; Obesity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motion-controlled video gaming (Experimental): Participants played motion-controlled video games that involved at least throwing, hitting, or dancing motions using a Wii or Xbox 360 console for one hour
  Interventions: Other: Motion-controlled video gaming
- Traditional video gaming (Active Comparator): Participants played traditional (handheld gamepad controller-based) video games using a Playstation 3 console for one hour
  Interventions: Other: Traditional video gaming
- Television watching (Active Comparator): Participants watched television via Netflix instant streaming for one hour
  Interventions: Other: Television watching

INTERVENTIONS:
Other: Motion-controlled video gaming — Play of motion-controlled video games for one hour
  Arms: Motion-controlled video gaming
Other: Traditional video gaming — Participants played traditional video games for one hour
  Arms: Traditional video gaming
Other: Television watching — Participants watched television for one hour
  Arms: Television watching

SUMMARY:
The purpose of this study is to determine whether playing motion-controlled video games produces low caloric intake and higher caloric expenditure than watching TV or playing traditional video games.

DETAILED DESCRIPTION:
The purpose of this study is to investigate differences in behaviors and emotions during TV watching and video game playing. Participants will be randomized to either watch TV, play traditional button-based video games, or play motion-based video games for one hour while palatable snack foods and sugar-sweetened beverages are provided within easy reaching distance. Both energy intake as well as energy expenditure during a one-hour period will be measured. All three conditions will be optimized to resemble typical in-home conditions as much as possible.

An additional goal of this study is to provide insight into the possible pathways by which TV and video games differentially affect intake and expenditure. Distraction from the real world (also called presence or engagement) will be analyzed to determine if a) these variables differ across groups and b) if these variables explain differences in energy intake and/or expenditure. The TV group will watch TV shows using Netflix streaming service, which will allow them to choose from a variety of popular shows without viewing commercials. As the investigators are primarily interested in satiety and hand occupation effects, the lack of commercials will allow us to eliminate food advertisements as a causal factor.

Finally, the third major goal of the study is to investigate how young adults choose screen-based media. In the two video game arms, participants will be allowed to choose to play any of 10 provided games, and in the TV group, participants will be able to choose from hundreds of options. Choices of game/program, time spent on each game/program, and psychological reactions to each game will be measured and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35 years old

Exclusion Criteria:

* Not at least a novice video game played (defined as having played games once or twice within the last year)
* Has pre-existing medical condition that precludes physical activity
* Is unable to find transportation to the study center
* Does not agree to be videotaped during the experiment
* Does not agree or is unable to fast for two hours prior to the experiment
* Is pregnant or nursing
* Weighs more than 300 pounds (required by one of the game controllers)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Energy intake | One-hour study period
  Energy intake was measured by weighing available food and beverage containers before and after one-hour period in which participants watched TV/played video games, then calculating the differences in weights

SECONDARY OUTCOMES:
Energy expenditure | One-hour study period
  Energy expenditure was measured using a Sense Wear Pro armband, which uses accelerometry and galvanic skin response to estimate metabolic equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Lyons, PhD, MPH, Principal Investigator — University of Texas
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Lyons EJ, Tate DF, Ward DS, Wang X. Energy intake and expenditure during sedentary screen time and motion-controlled video gaming. Am J Clin Nutr. 2012 Aug;96(2):234-9. doi: 10.3945/ajcn.111.028423. Epub 2012 Jul 3. PMID 22760571